CLINICAL TRIAL: NCT03288129
Title: Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of Perampanel as Monotherapy or First Adjunctive Therapy in Subjects With Partial Onset Seizures With or Without Secondarily Generalized Seizures or With Primary Generalized Tonic-Clonic Seizures
Brief Title: Study to Evaluate the Efficacy and Safety of Perampanel as Monotherapy or First Adjunctive Therapy in Subjects With Partial Onset Seizures With or Without Secondarily Generalized Seizures or With Primary Generalized Tonic-Clonic Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-G000-410; 2017-001180-20 (EudraCT Number)
Record Dates: First submitted 2017-09-13; First posted 2017-09-19 (Actual); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-04

CONDITIONS: Partial Onset Seizures; Secondarily Generalized Seizures; Primary Generalized Tonic-Clonic Seizures
Keywords: monotherapy; adjunctive therapy; open-label; multicenter
MeSH Terms: interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Perampanel (Experimental): Perampanel will be administered orally once daily (QD) at bedtime. At the beginning of the Titration Period, oral perampanel will start at a dose of 2 milligrams (mg) QD. Doses of perampanel will then be up titrated in increments of 2 mg at no less than 2-week intervals according to the investigator's judgment. At the 4 mg dose, the investigator will confirm whether further dose escalation is needed based on participant response and tolerability. The investigator may adjust dosing further or leave the participant at 4 mg. The maximum dose is 12 mg. During the 39-week Maintenance Period, participants will continue to receive the perampanel dose level that was administered at the end of the Titration Period.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — film-coated tablets
  Other Names: Fycompa; E2007

SUMMARY:
This study will assess the retention rate of perampanel when given as monotherapy or first adjunctive therapy in participants with partial-onset seizures or primary generalized tonic clonic seizures. The study consists of 4 periods: a Screening Period (to start no earlier than 6 weeks before the first dose of study drug), a Titration Period (up to 13 weeks), a Maintenance Period (39 weeks), and a Follow-Up Period (4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Participants will be male or female and no younger than 4 years of age and be able to swallow perampanel tablets.
* Participants must have a diagnosis of epilepsy with POS with or without SGS or with PGTCS. Either of the following must have occurred to support an epilepsy diagnosis:

  1. At least two unprovoked (or reflex) seizures occurring greater than 24 hours apart
  2. One unprovoked (or reflex) seizure with Electroencephalography (EEG) evidence of seizures
* Participants who receive perampanel as a first adjunctive therapy must currently have been treated with stable doses of monotherapy with an anti-epileptic drug (AED) for 8 weeks prior to Visit 2 (Week 0), have not previously received adjunctive AED treatment, and must, in the investigator's judgement, be in need of initial adjunctive therapy after failure to control seizures with AED monotherapy, at the optimal dose and duration.
* Participants who receive perampanel as monotherapy, who were newly diagnosed (treatment naïve), following the defined diagnosis of epilepsy.
* Participants who are currently receiving monotherapy treatment may receive perampanel as monotherapy if, in the investigator's judgment, the participant may benefit from a change in monotherapy treatment. Participants must not have previously received adjunctive AED treatment.
* If antidepressants or antianxiety drugs are used, participants must be on a stable dose regimen of these drugs during the 8 weeks before Visit 2 (Week 0).

Exclusion Criteria:

* Participants should not have previously received or currently be receiving perampanel.
* Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta human chorionic gonadotropin [β-hCG] or hCG test with a minimum sensitivity of 25 International Units per liter [IU/L] or equivalent units of β-hCG or hCG); a separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
* Females of childbearing potential who:

  * Within 28 days before study entry, did not use a highly effective method of contraception, which includes any of the following:

    * Total abstinence (if it is their preferred and usual lifestyle)
    * An intrauterine device or intrauterine hormone-releasing system
    * An oral contraceptive (with additional barrier method if using contraceptive containing levonorgestrel); participant must be on a stable dose of the same oral contraceptive product for at least 28 days before dosing and throughout the study and for 28 days after study drug discontinuation
    * Have a vasectomized partner with confirmed azoospermia
  * Do not agree to use a highly effective method of contraception (as described above) throughout the entire study period and for 28 days after study drug discontinuation For sites outside of the European Union, it is permissible that if a highly effective method of contraception is not appropriate or acceptable to the participant, then the participant must agree to use a medically acceptable method of contraception, i.e, double barrier methods of contraception such as condom plus diaphragm or cervical/vault cap with spermicide.

NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).

* Presence of or previous history of Lennox-Gastaut syndrome
* Presence of non-motor simple partial seizures only
* A history of status epilepticus within 1 year before Screening Visit (Visit 1)
* Participants on antipsychotics or who have psychotic disorder(s) or unstable recurrent affective disorder(s) with a history of attempted suicide within 1 year before Screening Visit (Visit 1)
* Presence of a progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors
* Concomitant use of barbiturates (except for seizure control indication and premedication for electroencephalogram) and benzodiazepines (except for seizure control indication) within 8 weeks prior to Visit 2 (Week 0)
* Use of intermittent rescue benzodiazepines (i.e, 1 to 2 doses over a 24-hour period is considered a one time rescue) 2 or more times in the 8-week period prior to Visit 2 (Week 0)
* Severe renal insufficiency (defined by estimated glomerular filtration rate of < 30 milliliters per minute [mL/min]) or participants who receive hemodialysis
* Evidence of clinically significant disease (eg, cardiac, respiratory, gastrointestinal, renal disease, hepatic disease) that in the opinion of the investigator(s) could affect the participant's safety or study conduct NOTE: Stable elevation of liver enzymes, alanine aminotransferase and aspartate aminotransferase due to concomitant medication(s) will be allowed if they are less than 3 times the upper limits of normal.
* Hypersensitivity to perampanel or any excipients
* Participants with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
* Participants who are participating in other interventional clinical trial
* Participant who are judged to have inadequate cognitive ability for participation in the study (intelligence quotient < 80 or investigator judgment)
* Any suicidal ideation with intent with or without a plan, at the time of or within 6 months of screening, as indicated by answering "Yes" to questions 4 and 5 on the Suicidal Ideation section of the Columbia Suicide Severity Rating Scale (C-SSRS)
* Any lifetime suicidal behavior based on the C-SSRS
* Concomitant use of any form of cannabidiol (CBD)
* Planned brain surgery during study participation

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - The Board of Trustees of the University of Alabama for the University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - Arkansas Epilepsy Program, Little Rock, Arkansas
  - UCSD Epilepsy Center, La Jolla, California
  - Stanford Medical Center, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - Baptist Health, Nemours Children's Specialty Care, Jacksonville, Florida
  - RUSH University Medical Center, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - The Regents of The University of Michigan, Ann Arbor, Michigan
  - Michigan State University, East Lansing, Michigan
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - JFK Medical Center, Edison, New Jersey
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - UNM Health Providers, Albuquerque, New Mexico
  - Mount Sinai Medical Center, New York, New York
  - Duke Neurology, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 14 investigative sites in the United States from 23 August 2017 to 27 April 2021.
Pre-assignment Details: A total of 68 participants were screened, of which 54 were treated with perampanel.
Groups:
- Perampanel 12 mg: During the Titration Period, participants received perampanel 2 milligrams per day (mg/day) and were up-titrated in no less than 2-week intervals in increments of 2 milligram (mg) up to 12 mg were allowed based on the participants response and tolerability and at the investigator's judgment. Upon entering the Maintenance Period, participants received the last dose they achieved at the end of the Titration Period and continued receiving this dose once daily for up to 39 weeks.
Period: Overall Study
Arm/Group | Perampanel 12 mg
Started | 54
Completed | 32
Not Completed | 22
Not completed — Adverse Event | 10
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 3
Not completed — Withdrawal of consent/assent | 1
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.
Groups:
- Perampanel 12 mg: During the Titration Period, participants received perampanel 2 mg/day and were up-titrated in no less than 2-week intervals in increments of 2 mg up to 12 mg were allowed based on the participants response and tolerability and at the investigator's judgment. Upon entering the Maintenance Period, participants received the last dose they achieved at the end of the Titration Period and continued receiving this dose once daily for up to 39 weeks.
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (17.32) [lower limit 17.32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 42
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Remaining on Perampanel Treatment at 3 Months After the Initiation of Treatment
Description: The retention rate was defined as the percentage of participants remaining on perampanel treatment at 3 months after the initiation of treatment.
Time Frame: Month 3
Population: The Safety Analysis Set included participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 54
percentage of participants | 85.2

2. Primary Outcome: Percentage of Participants Remaining on Perampanel Treatment at 6 Months After the Initiation of Treatment
Description: The retention rate was defined as the percentage of participants remaining on perampanel treatment at 6 months after the initiation of treatment.
Time Frame: Month 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 54
percentage of participants | 68.5

3. Primary Outcome: Percentage of Participants Remaining on Perampanel Treatment at 9 Months After the Initiation of Treatment
Description: The retention rate was defined as the percentage of participants remaining on perampanel treatment at 9 months after the initiation of treatment.
Time Frame: Month 9
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 54
percentage of participants | 63.0

4. Primary Outcome: Percentage of Participants Remaining on Perampanel Treatment at 12 Months After the Initiation of Treatment
Description: The retention rate was defined as the percentage of participants remaining on perampanel treatment at 12 months after the initiation of treatment.
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 54
percentage of participants | 51.9

5. Secondary Outcome: Percentage of Participants Who Achieved Seizure-free Status During the Maintenance Period
Description: Seizure-free status was defined as no incidence of seizure during the entire maintenance period. Partial seizures: when abnormal electrical activity begins in only one part of brain include (1) simple partial seizures: participants does not lose consciousness may experience muscle jerking or stiffening, (2) complex partial seizures: participant loses awareness. SGS: disturbances that spread to both sides of brain after partial seizure has already begun and happen when burst of electrical activity in limited area (the partial seizure) spreads throughout brain. PGTCS: disturbances in functioning of both sides of brain that caused by electrical signals spreading through brain inappropriately.
Time Frame: Up to 39 weeks of Maintenance Period
Population: The Full Analysis Set (FAS) included participants who received at least 1 dose of study drug and had at least 1 postdose seizure measurement. Here "overall number of participants analyzed" signifies participants those who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 52
percentage of participants | 19.2

6. Secondary Outcome: Percentage of Participants Who Achieved 3-month Seizure-free Status During the Maintenance Period
Description: Seizure-free status was defined as no incidence of seizure at 3 months during the Maintenance Period. Partial seizures: when abnormal electrical activity begins in only one part of brain include (1) simple partial seizures: participant does not lose consciousness may experience muscle jerking or stiffening, (2) complex partial seizures: participant loses awareness. SGS: disturbances that spread to both sides of brain after partial seizure has already begun and happen when burst of electrical activity in limited area (the partial seizure) spreads throughout brain. PGTCS: disturbances in functioning of both sides of brain that caused by electrical signals spreading through brain inappropriately.
Time Frame: Up to 3 months of Maintenance Period
Population: The FAS included participants who received at least 1 dose of study drug and had at least 1 postdose seizure measurement. Here "overall number of participants analyzed" signifies participants those who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 52
percentage of participants | 34.6

7. Secondary Outcome: Percentage of Participants Who Achieved 6-month Seizure-free Status During the Maintenance Period
Description: Seizure-free status was defined as no incidence of seizure at 6 months during Maintenance Period. Partial seizures: when abnormal electrical activity begins in only one part of brain include (1) simple partial seizures: participant does not lose consciousness may experience muscle jerking or stiffening, (2) complex partial seizures: participant loses awareness. SGS: disturbances that spread to both sides of brain after partial seizure has already begun and happen when burst of electrical activity in limited area (the partial seizure) spreads throughout brain. PGTCS: disturbances in functioning of both sides of brain that caused by electrical signals spreading through brain inappropriately.
Time Frame: Up to 6 months of Maintenance Period
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 52
percentage of participants | 23.1

8. Secondary Outcome: Percentage of Participants Who Received Perampanel as a First Adjunctive Therapy and Converted to Perampanel Monotherapy
Description: Percentage of participants who received perampanel as a first adjunctive therapy and converted to perampanel monotherapy were reported.
Time Frame: Up to 52 weeks
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 52
percentage of participants | 28.8

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAE)
Description: A TEAE was defined as an adverse event (AE) that emerged during treatment, having been absent at pretreatment (Baseline) or reemerged during treatment, having been present at pretreatment (Baseline) but stopped before treatment, or worsened in severity during treatment relative to the pretreatment state, when the AE was continuous.
Time Frame: From date of first administration of study drug up to 28 days after last dose of study drug (up to 56 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 54
Participants | 48

10. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (SAE)
Description: A SAE was defined as any untoward medical occurrence that at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect. A TEAE was defined as an event that emerges during treatment having been absent pre-treatment, or worsens relative to the pre-treatment state.
Time Frame: From date of first administration of study drug up to 28 days after last dose of study drug (up to 56 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 54
Participants | 4

ADVERSE EVENTS:
Time Frame: From date of first administration of study drug up to 28 days after last dose of study drug (up to 56 weeks)
Arm/Group | Perampanel 12 mg
All-Cause Mortality (participants affected / at risk) | 1/54
Serious Adverse Events (participants affected / at risk) | 4/54
Other Adverse Events (participants affected / at risk) | 47/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perampanel 12 mg (N=54)
Sudden unexplained death in epilepsy (General disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perampanel 12 mg (N=54)
Nausea (Gastrointestinal disorders) | 4 (7)
Vomiting (Gastrointestinal disorders) | 6 (6)
Fatigue (General disorders) | 9 (12)
Upper respiratory tract infection (Infections and infestations) | 3 (4)
Nasopharyngitis (Infections and infestations) | 5 (6)
Balance disorder (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 15 (19)
Headache (Nervous system disorders) | 5 (5)
Memory impairment (Nervous system disorders) | 3 (3)
Somnolence (Nervous system disorders) | 8 (10)
Aggression (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 3 (3)
Irritability (Psychiatric disorders) | 5 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Ear infection (Infections and infestations) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT03288129/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT03288129/SAP_001.pdf